CLINICAL TRIAL: NCT00995085
Title: Efficacy Study of Metadoxine SR Formulation in ADHD Subjects
Brief Title: Efficacy Study of Metadoxine SR Formulation in Attention Deficit Hyperactivity Disorder (ADHD) Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alcobra Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0012-09-GEH
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2011-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; ADD; TOVA; METADOXINE
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — metadoxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metadoxine SR (Experimental): Metadoxine is a pyrolate salt of Pyridoxine
  Interventions: Drug: Extended Release Metadoxine

INTERVENTIONS:
Drug: Extended Release Metadoxine — one oral 1400mg dose (2 tablets)
  Other Names: Metadoxine, Metadoxil

SUMMARY:
This clinical study is designed to evaluate the safety and tolerability of a single oral administration of a Metadoxine slow release formulation to subjects diagnosed as having ADHD. Study also assess cognitive effects of such drug administration.

DETAILED DESCRIPTION:
Primary outcome measure is the safety and tolerability of study drug after a single dosing.

Additional outcomes include commission error rate from the TOVA test. The result is measured as standard score in % compared to the values of the normal population.

Exploratory outcome measures include:

1. TOVA measures like response time , variability, omissions etc.
2. Subtests from Wechsler: digit memory, digit-number signs etc

ELIGIBILITY:
Inclusion Criteria:

* age 18-45
* diagnosed as ADHD

Exclusion Criteria:

* PDD patients
* head injured patients
* patients suffering from heart, lung, liver, kidney, intestinal, endocrine an neurological diseases and patients who are sensitive to vitamin B

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Manor, MD, Principal Investigator — Geha MC, Israel
Locations (1):
- ADHD Unit, Geha MHC, Israel, Petah Tikva, Israel

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metadoxine SR
Started | 43
Completed | 38
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Metadoxine SR
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 25
Region of Enrollment [Number; unit: participants]
  Israel | 43

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Subjects were evaluated for general safety and tolerablity measures, including number of AEs and AEs related (possibly or likely) to study drug
Time Frame: 24 hours after drug adminstration
Measure: Number; unit: events
Arm/Group | Metadoxine SR
Number analyzed (Participants) | 43
events | 2

ADVERSE EVENTS:
Arm/Group | Metadoxine SR
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 2/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metadoxine SR (N=38)
Tiredness (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less